CLINICAL TRIAL: NCT05432752
Title: Use of the Concussion Pen in Evaluating Ocular-motor Function in the Concussed and Non-concussed Populations Ages 11 to 18 Years Old.
Brief Title: Concussion Pen Screening Tool
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Mercy Hospital Kansas City (Other)
Responsible Party: Principal Investigator, Andrea Thorne, Principal Investigator, PT, Children's Mercy Hospital Kansas City
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: STUDY00002250
Record Dates: First submitted 2022-06-21; First posted 2022-06-27 (Actual); Last update posted 2023-03-02 (Actual); Status verified 2023-02

CONDITIONS: Fixation, Ocular; Brain Concussion
Keywords: Ocular motor function; Concussion
MeSH Terms: conditions — Brain Concussion

STUDY DESIGN:
Intervention Model Description: All subjects will undergo clinical evaluation for concussion and will also be evaluated using the Concussion Pen. All subjects (both controls and concussion patients) will undergo all eye tracking measurements. Randomization to being evaluated using clinical care first then the Concussion Pen and vice versa will be utilized.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Concussed Subjects (Experimental): Subjects with known history of concussion will be evaluated using current clinical evaluation and also using the Concussion Pen.
  Interventions: Device: Concussion Pen
- Non-Concussed Subjects (Experimental): Subjects with no known history of concussion will be evaluated using current clinical evaluation for a concussion and also using the Concussion Pen.
  Interventions: Device: Concussion Pen

INTERVENTIONS:
Device: Concussion Pen — Device will measure the distance from the eye to the Concussion Pen for ocular motor functions.

SUMMARY:
To compare the use of the Concussion Pen to current clinical care practice. This will be a prospective study of a maximum of 24 subjects, with a goal enrollment of 20 subjects (10 in each cohort). All subjects will undergo clinical evaluation for concussion and will also be evaluated using the Concussion Pen. Randomization to being evaluated using clinical care first then the Concussion Pen and vice versa will be utilized. This randomization will help to control for evaluation fatigue on the part of study participants.

DETAILED DESCRIPTION:
This will be a prospective study of a maximum of 24 subjects, with a goal enrollment of 20 subjects (10 in each cohort). All subjects will undergo clinical evaluation for concussion and will also be evaluated using the Concussion Pen. All subjects (both controls and concussion patients) will undergo all eye tracking measurements. Randomization to being evaluated using clinical care first then the Concussion Pen and vice versa will be utilized.

This will be a multi-disciplinary team with members of Physical Therapy (PT)/ Occupational Therapy (OT), Medical Doctor (MD), Doctor of Osteopathic Medicine (DO), and Doctor of Philosophy(PhD)s who specialize in concussion assessment. This study will include a population of concussed patients as well as non-concussed patients (controls) who will be seen in CM clinics per standard of care.

ELIGIBILITY:
Inclusion Criteria:

Inclusion Criteria for both control and study cohorts, unless stated otherwise below

* Patients cognitively 11 to 18 years of age.
* Patients undergoing evaluation for concussion in Children's Mercy (CM) clinics for concussion population.
* Patients with a history of concussion at any previous point in time (no time limits to this date).
* Patients with no history of concussion and being seen at CM PT/OT for other diagnoses for control population.
* Patients able to give verbal assent or consent (dependent on patient cognitive age), and Legally Authorized Representatives (LAR)s able to give verbal parental permission.
* English-speaking families.

Exclusion Criteria:

* Patients not within the inclusion criteria as outlined above.
* Patients with congenital vestibular dysfunction will not be included.
* Patients diagnosed with dyslexia or Attention Deficit Hyperactive Disorder (ADHD) will not be included.
* Non-English-speaking families.
* Wards of the State will not be approached for this study.
* Patients with a previous diagnosis of strabismus or convergence insufficiency will be excluded.

Ages: 11 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 21 (Actual)
Dates: Start 2022-07-28 (Actual); Primary Completion 2023-01-25 (Actual); Study Completion 2023-01-25 (Actual)

PRIMARY OUTCOMES:
Concussion Pen versus Current Clinical Evaluation | 1 year
  Concussion Pen is able to determine concussed patients to the same level as current clinical evaluation.

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Thorne, PT, Principal Investigator — Children's Mercy Hospital Kansas City
Locations (1):
- Children's Mercy Hospital, Kansas City, Missouri, United States

IPD SHARING:
Plan to Share IPD: No